CLINICAL TRIAL: NCT04290546
Title: A Phase 1 Trial of CTLA-4 Inhibition, With or Without Cetuximab, and in Combination With Memory-like Natural Killer (NK) Cell Immune Cell Therapy in Advanced Head & Neck Cancer
Brief Title: CIML NK Cell in Head & Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Altor BioScience (Industry); Bristol-Myers Squibb (Industry); Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-505
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of the Head and Neck; Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ALT-803; Ipilimumab; Immune Checkpoint Inhibitors; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort I without Ipilimumab Lead in (Experimental): Haploidentical donor derived CIML NK cell infusion with subcutaneous N-803 for eligible patients with platinum-refractory and immune checkpoint blockade-refractory, advanced head and neck squamous cell carcinoma (Cohort 1)
  * CIML NK cell infusion (Dose 0 or -1) infused on Day 0.
  * Interleukin-15 Superagonist dosed at 15 mcg/kg subcutaneously every 21 days for 4 total doses (a cycle being every 21-days, so 4 cycles).
  Interventions: Drug: Interleukin-15 Superagonist (N-803); Biological: CIML NK cell Infusion
- Cohort 2 with Ipilimumab Lead In (Experimental): Cohort 2 treated with an ipilimumab lead-in prior to CIML NK cell infusion after safety is established with the NK cell and N-803 treatments alone.
  * Participants in the ipilimumab subgroup (Cohort 2) will receive a single dose of lead-in ipilimumab via iv per protocol determined dose followed by lymphodepleting chemotherapy on Day -6 for a total of 5-days, prior to receiving CIML NK cell infusion.
  * CIML NK cell infusion-Highest Dosed per cohort 1, infused on day 0
  * Interleukin-15 Superagonist (N-803) Administration
    -- dosed at 15 mcg/kg subcutaneously every 21 days for 4 total doses (a cycle being every 21-days, so 4 cycles).
  * Cohort 2 will receive the highest number of CIML NK cells that is still considered safe and ipilimumab.
  Interventions: Drug: Interleukin-15 Superagonist (N-803); Biological: CIML NK cell Infusion; Drug: Ipilimumab
- Cohort 3 with Cetuximab Infusions (Experimental): Cohort 3 treated with CIML NK cell infusion after safety is established with the NK cell and N-803 treatments alone, followed by cetuximab infusions.
  * - Participants in cetuximab subgroup (Cohort 3) will receive lymphodepleting chemotherapy on Day -6 for a total of 5-days, prior to receiving CIML NK cell infusion.
  * CIML NK cell infusion-Highest Dosed per cohort 1, infused on day 0
  * Interleukin-15 Superagonist (N-803) Administration
    -- dosed at 15 mcg/kg subcutaneously every 21 days for 4 total doses (a cycle being every 21-days, so 4 cycles).
  * Cetuximab Administration
    --dosed at 500mg/m2 IV over 120 minutes for the first dose, then over 60 minutes for subsequent doses. This will be infused every 14 days for 8 doses started on day +15.
  * Cohort 3 will receive the highest number of CIML NK cells that is still considered safe and ipilimumab.
  Interventions: Drug: Interleukin-15 Superagonist (N-803); Biological: CIML NK cell Infusion; Drug: Cetuximab

INTERVENTIONS:
Drug: Interleukin-15 Superagonist (N-803) — -- Starting the day after (Cycle 1, Day +1) CIML NK-enriched cell infusion, at least 12 hours after CIML NK cell infusion is completed and up to 48 hours after CIML NK cell infusion, each participant will receive N-803 dosed at 15 mcg/kg subcutaneously every 21 days for 4 total doses (a cycle being every 21-days, so 4 cycles).
  N-803 dosed at 15 mcg/kg subcutaneously every 21 days for 4 total doses (a cycle being every 21-days, so 4 cycles) for cohorts 1 and 2, and 6 total doses in cohort 3. The dose should be calculated based on body weight at study entry, and recalculated only if greater than 10% change in weight.
Biological: CIML NK cell Infusion — (Dose 0 or -1) infused on Day 0
  Other Names: cytokine induced memory-like natural killer
Drug: Ipilimumab — single dose of lead-in ipilimumab via iv per protocol determined dose
  Other Names: CTLA-4 inhibitor
  Arms: Cohort 2 with Ipilimumab Lead In
Drug: Cetuximab — Starting day +15, every 14 days for 8 total doses via IV per protocol
  Other Names: EGFR inhibitor
  Arms: Cohort 3 with Cetuximab Infusions

SUMMARY:
This research study is evaluating the safety and efficacy of a combination drug and biologic therapy in patients with advanced head and neck cancer.

This research study involves the following drugs and biologics:

* CIML NK donor cells
* IL-15 superagonist
* Ipilimumab
* Cetuximab

DETAILED DESCRIPTION:
This is a three-part, non randomized, open label, single site Phase 1 study. The purpose of this research study is to obtain information on the safety and effectiveness of this combination of study drugs to treat advanced head and neck. The experimental combination therapy in this study involves CIML NK cells from a haploidentical donor (meaning cells from another person with similar immune proteins), IL-15, participants in cohort 2 will also receive ipilimumab, and participants in cohort 3 will receive cetuximab. CIML NK cells are an allogeneic cell product derived from qualified donor natural killer (NK) cells that have been bathed in special proteins to help to identify and treat certain advanced cancers.

- Participants who fulfill eligibility criteria will be entered into the trial CTLA-4 Inhibition in Combination with Memory-like Natural Killer (NK) Cell Immune Cell Therapy in Advanced Head & Neck Cancer.

The study consists of 3 parts:

* Cohort 1 CIML NK cells without ipilimumab
* The investigators are looking the highest dose of the study intervention that can be administered safely without severe or unmanageable side effects in participants that have advanced head and neck cancer, not everyone who participates in this research study will receive the same dose of the study intervention. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated
* Cohort 2 participants will be treated at the respective dose (at or below the Maximum Tolerated Dose), as determined during Cohort plus a lead-in dose of ipilimumab
* Cohort 3 participants will be treated at the respective dose (at or below the Maximum Tolerated Dose), as determined during Cohort plus infusions of cetuximab
* It is expected that about 25 people will take part in this research study.

This research study is a Phase I clinical trial, which tests the safety of investigational drugs and tries to define the appropriate dose of the investigational drugs to use for further studies.

"Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved CIML NK cells as treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved IL-15 as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved ipilimumab for your specific disease but it has been approved for other uses.

The U.S. Food and Drug Administration (FDA) has approved cetuximab for your specific disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, recurrent or metastatic squamous cell carcinoma of the head neck (including oral cavity, oropharynx, larynx, hypopharynx, paranasal sinuses) or salivary gland carcinoma (including adenoid cystic carcinoma and non-adenoid cystic carcinoma histologies)
* Any HPV status or smoking history is permitted. Oropharyngeal cancer patients are required to undergo HPV testing with p16 immunohistochemistry and/or confirmatory HPV PCR or ISH testing
* Available haploidentical donor that is willing and eligible for non-mobilized collection
* Prior exposure to a platinum-containing regimen (either in the definitive or advanced, recurrent/metastatic setting) and exposure to a PD-1/L1 inhibitor is required for SCCHN patients only
* Age 18 years or older
* ECOG performance status ≤ 2 (see Appendix A).
* No systemic corticosteroid therapy (≤ 10 mg of prednisone or equivalent dose of systemic steroids for non-autoimmune indications for at least 4 weeks prior to NK cell infusion).
* Ability to understand and the willingness to sign a written informed consent document.
* Negative pregnancy test for women of childbearing potential only. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.
* The effects of CIML NK cells and N-803 on the developing human fetus are unknown.

For this reason, WOCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for up to 26 weeks after the last dose of all investigational products (up to 16 weeks after the last N-803 dose), in such a manner that the risk of pregnancy is minimized. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

* Willing to provide blood and tissue from diagnostic biopsy and at the time of surgery
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥ 2,500/mcL
  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 90,000/mcL
  * total bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3x institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * Oxygen saturation: ≥ 90% on room air
  * Left ventricular ejection fraction (cardiac function) > 40%

Exclusion Criteria:

* Patients with nasopharyngeal carcinoma are not eligible
* Participants who have had anti-tumor chemotherapy or other investigational agents within 2 weeks prior to cell infusion (6 weeks for nitrosoureas or mitomycin C), or immunotherapy within 3 weeks prior, or those who have not recovered from adverse events due to agents administered more than 3 weeks prior.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to N-803 or other agents used in study.
* Solid organ transplant (allograft) recipients.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [Wegener's granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain- Barre syndrome and myasthenia gravis). Patients with Hashimoto thyroiditis are eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and N-803 and with the potential for teratogenic or abortifacient effects by fludarabine/cyclophosphamide chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and N-803, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Individuals with active uncontrolled hepatitis B or C are ineligible as they are at high-risk of lethal treatment-related hepatotoxicity in the setting of marrow suppression.
* Known non-infectious pneumonitis or any history of interstitial lung disease.
* Receipt of a live vaccine within 30 days of start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Rate of Dose Limiting Toxicity | first dose of study treatment up to 100 days
  All patients receiving any dose of study treatment will be evaluated for safety. DLTs overall and by dose level will be reported as proportions with 90% exact binomial confidence intervals.

SECONDARY OUTCOMES:
objective response rate (ORR) | 12 weeks
  reported as proportions with 90% exact binomial confidence intervals for all patients and by dose level
complete response (CR) rate | 12 weeks
  reported as proportions with 90% exact binomial confidence intervals for all patients and by dose level
disease-free survival (DFS) | 1 year
  Kaplan and Meier
overall survival (OS) at 1-year following infusion | 1 year
  Kaplan and Meier

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Shapiro RM, Sheffer M, Booker MA, Tolstorukov MY, Birch GC, Sade-Feldman M, Fang J, Li S, Lu W, Ansuinelli M, Dulery R, Tarannum M, Baginska J, Dwivedi N, Kothari A, Penter L, Abdulhamid YZ, Kaplan IE, Khanhlinh D, Uppaluri R, Redd RA, Nikiforow S, Koreth J, Ritz J, Wu CJ, Soiffer RJ, Hanna GJ, Romee R. First-in-human evaluation of memory-like NK cells with an IL-15 super-agonist and CTLA-4 blockade in advanced head and neck cancer. J Hematol Oncol. 2025 Feb 14;18(1):17. doi: 10.1186/s13045-025-01669-3. PMID 39948608